CLINICAL TRIAL: NCT04083963
Title: BRE-01: Phase 2 Trial of Neoadjuvant Weekly Carboplatin Plus Paclitaxel Followed by Doxorubicin and Cyclophosphamide in Triple Negative Breast Cancer
Brief Title: Phase 2 Trial of Neoadjuvant Weekly Carboplatin Plus Paclitaxel in Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kent F. Hoskins, MD, Associate Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0550
Record Dates: First submitted 2019-08-21; First posted 2019-09-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Carboplatin; Paclitaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Carboplatin plus paclitaxel followed by doxorubicin and cyclophosphamide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Other): Low dose weekly carboplatin in combination with standard neoadjuvant chemotherapy
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Carboplatin — Low dose weekly carboplatin (AUC 2) will be combined with weekly paclitaxel for 12 weeks.
  Other Names: Paraplatin
Drug: Paclitaxel — Paclitaxel will be given weekly along with carboplatin for 12 weeks.
  Other Names: Taxol
Drug: Doxorubicin — Dose dense doxorubicin will be administered in combination with cyclophosphamide for 4 cycles after weekly carboplatin/paclitaxel.
  Other Names: Adriamycin
Drug: Cyclophosphamide — Does dense cyclophosphamide will be in combination with doxorubicin for 4 cycles after weekly carboplatin/paclitaxel.
  Other Names: Cytoxan

SUMMARY:
Nonrandomized, open label, single arm, Simon's two stage MinMax design trial of neoadjuvant weekly carboplatin plus paclitaxel, followed by doxorubicin and cyclophosphamide in patients with operable Triple Negative Breast Cancer (TNBC)

DETAILED DESCRIPTION:
This is a single arm, Phase 2, open label, Simon's two stage MinMax design trial to evaluate the safety and efficacy of weekly carboplatin in combination with standard neoadjuvant chemotherapy in subjects with previously untreated triple negative breast cancers who are candidates for potentially curative surgery.

Subjects will receive carboplatin (Area Under the Curve (AUC) 2 mg/mL/min) + paclitaxel (80 mg/m2) Carboplantin plus Paclitaxel (CbP) followed by doxorubicin and cyclophosphamide (AC). All subjects will receive CbP on Day 1 of 12 weekly cycles (Visits CbP1 - CbP12) via infusion during Chemotherapy Segment 1 as indicated in the Study Schema. Dose interruptions and dose modifications are allowed based upon tolerability and may extend Chemotherapy Segment 1 duration to a maximum of 16 weeks. Beginning with Chemotherapy Segment 2 all subjects will receive doxorubicin (60 mg/m2) and cyclophosphamide (600 mg/m2) on Day 1 of four 14-day cycles (Visits AC1 - AC4). For subjects who experience toxicities due to carboplatin, paclitaxel, doxorubicin or cyclophosphamide, the appropriate dose modifications or dosing delays should be managed according to Section 11.2. Dose modifications may result in the total duration of therapy being greater than the planned 24 weeks. The objective of this study is to determine efficacy and tolerability of low dose, weekly carboplatin in combination with weekly paclitaxel followed by standard doxorubicin/cyclophosphamide as neoadjuvant therapy for triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female ≥ 18 years of age at time of consent.
2. Histologically confirmed invasive breast carcinoma documented by core needle biopsy or incisional biopsy (excisional biopsy is not allowed). AJCC clinical stage T1c, N0-3 or cT1, N1-3 by physical exam or radiologic studies. Suspected involvement of regional lymph nodes based on physical exam or imaging studies must be confirmed cytologically/histologically.
3. Surgical excision of the primary breast tumor (partial mastectomy or total mastectomy) and ipsilateral axillary lymph node sampling (sentinel lymph node biopsy or axillary dissection) are planned following neoadjuvant chemotherapy.
4. Estrogen Receptor (ER)- and Progesterone Receptor (PR)-negative, and Human Epidermal Growth Factor Receptor (HER)2-negative (triple-negative) cancer of the breast.

   Triple-negative tumors are defined as:
   * ER- and PR-negative: less than or equal to 10% tumor staining by immunohistochemistry (IHC) according to local pathology assessment.
   * HER2-negative disease, defined as defined by ASCO/CAP guidelines [24]. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 within 28 days prior to study registration.
5. Life expectancy of 6 months or greater as determined by the treating physician.
6. Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 28 days prior to registration.

   System Hematological Leukocytes
   * 2,500/mm3 Platelet count
   * 100,000/mm3 Absolute Neutrophil Count (ANC)
   * 1,500/mm3 Hemoglobin (Hgb)
   * 9.5 g/dL Renal Creatinine/Calculated creatinine clearance (CrCl) Cr < 1.5 x upper limit of normal (ULN) or CrCl ≥ 50 mL/min using the Cockcroft-Gault formula Hepatic Bilirubin Bilirubin ≤ 1.5 × ULN. Subjects with Gilbert's syndrome may have a bilirubin > 1.5 × ULN, if no evidence of biliary obstruction exists Aspartate aminotransferase (AST)

     * 2.5 × ULN Alanine aminotransferase (ALT)
     * 2.5 × ULN
7. No evidence of distant metastases (M0 as per AJCC staging guidelines) Weekly Carboplatin for TNBC Confidential Protocol v.1.0, dated February 10, 2019 Page 19 of 64
8. Provided written informed consent and HIPAA authorization for release of personal health information, approved by an Institutional Review Board (IRB).
9. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
10. Women of childbearing potential (WOCP) must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required within 14 days of study registration. If the urine test cannot be confirmed as negative, a serum pregnancy test will be required.
11. Women of childbearing potential (WOCP) must be willing to use two effective methods of birth control such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence for the course of the study until 90 days after the last dose of study drug.

    NOTE: Women are considered to be of childbearing potential unless they are postmenopausal (≥45 years of age and has not had menses for greater than 12 consecutive months or bilateral oophorectomy) or surgically sterile (bilateral tubal ligation or hysterectomy) or not heterosexually active for the duration of the study and at least 60 days after the last dose of study drug.
12. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Active infection requiring systemic therapy.
2. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
3. Previous anti-cancer treatment (cytotoxic chemotherapy, immunotherapy, biologic therapy, radiotherapy directed towards the primary breast tumor and/or ipsilateral axillary lymph nodes or investigational agents) with therapeutic intent for the current breast cancer.
4. Previous treatment with carboplatin, paclitaxel, doxorubicin, or cyclophosphamide within the past 3 years.
5. Concurrent treatment with an ovarian hormonal replacement therapy or with hormonal agents such as raloxifene, tamoxifen or other selective estrogen receptor modulator (SERM). Subjects must have discontinued use of such agents prior to beginning study treatment.
6. A history of seizure within 6 months prior to study entry.
7. Pre-existing neuropathy from any cause in excess of Grade 1.
8. Treatment with any investigational drug within 14 days prior to registration or within 5 half-lives of the investigational product, whichever is longer.
9. Major surgery within 14 days prior to registration or has not recovered from major side effects
10. Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating Medical Oncologist.
11. Known history of AIDS (HIV testing is not mandatory). HIV-positive individuals on active HARRT therapy with virologic suppression (defined as an HIV-1 RNA level below the lower limit of detection of the assay used) within 90 days of study enrollment and a CD4 cell count >500 cells/mm3 on the most recent determination are eligible for the study.
12. History of myelodysplastic syndrome or acute myeloid leukemia.
13. Subjects with any of the following conditions:

    * History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 28 days prior to registration.
    * History of cerebrovascular accident (CVA) or transient ischemic attack within 6 months prior to registration.
    * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to registration.
    * Symptomatic congestive heart failure (New York Heart Association III-IV) or documented current left ventricular (LV) systolic dysfunction with left ventricular ejection fraction (LVEF) <50% on most recent assessment of LV function.
    * Clinically significant cardiac ventricular arrhythmias (e.g. sustained ventricular tachycardia/ventricular fibrillation) or high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block) unless a pacemaker is in place.
    * Any concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate subject participation in the clinical study or compromise compliance with the protocol.
14. Any condition that, in the opinion of the investigator, might jeopardize the safety of the patient or interfere with protocol compliance.
15. Any mental or medical condition that prevents the patient from giving informed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2026-09-27 (Estimated); Study Completion 2026-09-27 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | 30 months
  Defined as the absence of residual invasive carcinoma in the resected breast specimen and ipsilateral axillary lymph nodes following completion of neoadjuvant therapy (i.e., ypT0/Tis, ypN0 per the American joint Committee on Cancer staging system) in all subjects completing at least 1 cycle of study treatment (modified intent-to-treat population)

SECONDARY OUTCOMES:
Pathologic complete response rate in subjects completing protocol therapy. | 30 months
  Pathologic complete response rate Defined as the absence of residual invasive carcinoma in the resected breast specimen and ipsilateral axillary lymph nodes following completion of neoadjuvant therapy (i.e., ypT0/Tis, ypN0 per the American joint Committee on Cancer staging system) will be determined in the sub-group of subjects completing at least 75% of planned treatment cycles.
Residual Cancer Burden | 30 months
  The Residual Cancer Burden (RCB) class will be estimated from routine pathologic sections of the resected primary breast tumor and the regional lymph nodes after the completion of neoadjuvant therapy. RCB class 0 represents pCR, and class I represents minimal residual invasive disease. Class II and III represent significant residual disease. We will report the rate of achieving RCB class 0/1 vs. II/III.
Event-free survival (EFS) | 30 months
  Time from enrollment to any of the following: failure to undergo potentially curative surgery; onset of local, regional, or distant invasive recurrence of breast cancer following curative surgery; second primary invasive cancer in the breast or in another organ; or death from any cause.
Invasive disease-free survival (iDFS) | 30 months
  Time from enrollment to any of the following: development of invasive cancer in the ipsilateral breast or regional nodes, contralateral breast or regional nodes, distant metastases, or death from any cause
Distant disease-free survival (DDFS) | 30 months
  Time from enrollment to documentation of distant metastases or death from any cause
Overall survival (OS) | 30 months
  Time from enrollment to death from any cause
Clinical response to neoadjuvant chemotherapy | 30 months
  Defined as progressive disease, stable disease, partial response and complete response according to RECIST 1.1 criteria in the modified intent-to-treat population and participants completing at least 75% of protocol therapy
Breast conservation rate | 30 months
  The percentage of women undergoing adequate partial mastectomy as determined by treating physicians and achieving negative pathological surgical margins (no ink on tumor).
Treatment tolerability | 30 months
  Number of cycles delayed, deleted or requiring dose reduction; number of participants who fail to complete all planned courses of protocol therapy; number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Quality of life Measurement | 30 months
  Change in score on the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 quality of life survey. This 30-item survey uses a Likert scale with total scores ranging from 30-126, with increasing scores indicating worse quality of life. We will compare mean baseline scores to scores at the end of protocol therapy, and 3 and 12 months after completing all protocol therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Hoskins, M.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Chicago, Illinois, United States